CLINICAL TRIAL: NCT02518607
Title: A Single-centre, Double-blind, Placebo-controlled, Study in Healthy Men to Assess the Safety and Tolerability of Single and Repeated Ascending Doses of MGB-BP-3
Brief Title: Safety, Blood Levels and Effects of MGB-BP-3
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MGB Biopharma Limited (Industry)
Collaborators: Hammersmith Medicines Research (Other); Innovate UK (Other Government); Cambridge Regulatory Services (Unknown); Phases Clinical Research Limited (Unknown); Synlab Services (Unknown); Viapath (Unknown); Analytical Services International Limited (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14-019; 2015-000489-73 (EudraCT Number); MGB-BP-3-101 (Other: MGB Biopharma Limited)
Record Dates: First submitted 2015-07-29; First posted 2015-08-10 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Healthy
Keywords: Safety and Tolerability; Male Volunteers
MeSH Terms: interventions — MGB-BP-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (18):
- Group 1, Session 1, Active (Experimental): Lowest dose of SAD:
  MGB-BP-3, 250 mg liquid filled enterically coated capsule, single dose
  Interventions: Drug: MGB-BP-3
- Group 1, Session 2, Active (Experimental): Dose Escalation SAD:
  MGB-BP-3, 2X250 mg liquid filled enterically coated capsule, single dose
  Interventions: Drug: MGB-BP-3
- Group 1, Session 3, Active (Experimental): Dose Escalation SAD MGB-BP-3, 3X250 mg liquid filled enterically coated capsules, single dose
  Interventions: Drug: MGB-BP-3
- Group 2, Session 1, Active (Experimental): Dose Escalation SAD MGB-BP-3, 4X250 mg liquid filled enterically coated capsules, single dose
  Interventions: Drug: MGB-BP-3
- Group 2, Session 2, Active (Experimental): Dose Escalation SAD MGB-BP-3, 5X250 mg liquid filled enterically coated capsules, single dose
  Interventions: Drug: MGB-BP-3
- Group 2, Session 3, Active (Experimental): Dose Escalation SAD MGB-BP-3, 6X250 mg liquid filled enterically coated capsules, single dose
  Interventions: Drug: MGB-BP-3
- Group 3, Active (Experimental): Lowest dose of MAD MGB-BP-3, 2X250 mg liquid filled enterically coated capsules (AM/PM), multiple dose for 9 days and 1 single dose on Day 10
  Interventions: Drug: MGB-BP-3
- Group 4, Active (Experimental): Dose Escalation MAD MGB-BP-3, 4X250 mg liquid filled enterically coated capsules (2XAM/2XPM), multiple dose for 9 days and 1 single dose on Day 10
  Interventions: Drug: MGB-BP-3
- Group 5, Active (Experimental): Dose Escalation MAD MGB-BP-3, 8X250 mg liquid filled enterically coated capsules (3XAM/3XPM), multiple dose for 9 days and 1 single dose on Day 10
  Interventions: Drug: MGB-BP-3
- Group 1, Session 1, Placebo (Placebo Comparator): Lowest dose of SAD:
  Placebo, 1 liquid filled enterically coated capsule, single dose
  Interventions: Other: Placebo
- Group 1, Session 2, Placebo (Placebo Comparator): Placebo, 2 liquid filled enterically coated capsules, single dose
  Interventions: Other: Placebo
- Group 1, Session 3, Placebo (Placebo Comparator): Placebo, 3 liquid filled enterically coated capsules, single dose
  Interventions: Other: Placebo
- Group 2, Session 1, Placebo (Placebo Comparator): Placebo, 4 liquid filled enterically coated capsules, single dose
  Interventions: Other: Placebo
- Group 2, Session 2, Placebo (Placebo Comparator): Placebo, 5 liquid filled enterically coated capsules, single dose
  Interventions: Other: Placebo
- Group 2, Session 3, Placebo (Placebo Comparator): Placebo, 6 liquid filled enterically coated capsules, single dose
  Interventions: Other: Placebo
- Group 3, Placebo (Placebo Comparator): Placebo 2 liquid filled enterically coated capsules (AM/PM), multiple dose for 9 days and 1 single dose on Day 10
  Interventions: Other: Placebo
- Group 4, Placebo (Placebo Comparator): Placebo 4 liquid filled enterically coated capsules (2XAM/2XPM), multiple dose for 9 days and 1 single dose on Day 10
  Interventions: Other: Placebo
- Group 5, Placebo (Placebo Comparator): Placebo 8 liquid filled enterically coated capsules (3XAM/3XPM), multiple dose for 9 days and 1 single dose on Day 10
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: MGB-BP-3 — Treatment of CDI
  Other Names: MGB-BP-3-101
  Arms: Group 1, Session 1, Active; Group 1, Session 2, Active; Group 1, Session 3, Active; Group 2, Session 1, Active; Group 2, Session 2, Active; Group 2, Session 3, Active; Group 3, Active; Group 4, Active; Group 5, Active
Other: Placebo — Placebo
  Arms: Group 1, Session 1, Placebo; Group 1, Session 2, Placebo; Group 1, Session 3, Placebo; Group 2, Session 1, Placebo; Group 2, Session 2, Placebo; Group 2, Session 3, Placebo; Group 3, Placebo; Group 4, Placebo; Group 5, Placebo

SUMMARY:
This study is to assess the safety and tolerability aspects of oral MGB-BP-3, a treatment for Clostridium difficile infections.

DETAILED DESCRIPTION:
Short Title: Safety, blood levels and effects of MGB-BP-3

Trial medication MGB-BP-3 is a new class of antibacterial agent that binds selectively to the bacterial DNA minor groove and possesses strong bactericidal in vitro and in vivo activity against Clostridium difficile (C. difficile). In addition to its activity against C. difficile MGB-BP-3 has very strong activity against all other Gram-positive bacteria tested, including susceptible and resistant Staphylococcus aureus, Streptococcus and Enterococcus.

MGB-BP-3 is being developed for the treatment of C. difficile infections (CDI).

Objectives Primary: To assess the safety and tolerability of single and repeated oral doses of MGB-BP-3 in healthy men Secondary: To assess the pharmacokinetics (PK) of single and repeated oral doses of MGB-BP-3 in healthy men

Type of trial This trial will be done in 2 parts, as follows. Part A: Phase I, double-blind, randomised, placebo-controlled, crossover, single ascending-dose trial in healthy men.

Part B: Phase I, double-blind, randomised, placebo-controlled, sequential-group, repeated ascending-dose trial in healthy men.

Trial population Total up to 40 healthy men (excluding replacement subjects): 16 subjects in Part A and 24 subjects in Part B.

Age 18-45 years Principal inclusion criteria Normotensive male, with a body mass index (BMI) of 18.0-30.9 kg/m2; deemed healthy on the basis of a clinical history, physical examination, electrocardiogram (ECG), vital signs, and laboratory tests of blood and urine; willing to use reliable contraception; able to give fully informed written consent.

Principal exclusion criteria Positive tests for hepatitis B & C, HIV; severe adverse reaction to any drug; drug or alcohol abuse; smoke more than 5 cigarettes (or use of equivalent tobacco or nicotine products) daily; over-the-counter medication within previous 7 days (with the exception of paracetamol), or prescribed medication during previous 28 days; participation in other clinical trials of unlicensed medicines, or loss of more than 400 mL blood, within the previous 3 months; vital signs outside the acceptable range; clinically relevant abnormal findings at the screening assessment; acute or chronic illness; clinically relevant abnormal medical history or concurrent medical condition; possibility that volunteer will not cooperate.

Trial design and methods Part A Part A is a randomised, double-blind, placebo-controlled, cross-over, single ascending-dose trial in 16 healthy men. Subjects will be enrolled in 2 groups of 8 (Groups 1 and 2). Each subject will have 3 study sessions - they will receive a single oral dose of MGB-BP-3 in up to 3 study sessions; 6 volunteers will receive matching placebo in 1 study session.

So, at each dose level, 6 subjects will be randomised to receive MGB-BP-3 and 2 subjects will be randomised to receive placebo.

There will be a washout period of at least 4 days between doses for each subject, and an interval of at least 6 days between the last dose in Group 1 and the first dose in Group 2.

The investigator and sponsor will review the safety and tolerability data for each dose level before increasing the dose. The dose will only be escalated if the safety and tolerability of the previous dose level are acceptable. The planned dose level may be changed, based on emerging safety and tolerability data - a dose level may be repeated or a lower dose tested. The maximum dose tested will not exceed 2000 mg MGB-BP-3, which is 2-fold lower than the NOAEL (no observed adverse effect level) in male dog.

Because MGB-BP-3 has never been given to humans before, the first dose level will be staggered: 2 leading subjects will be dosed no later than the day before the remaining subjects in the group are dosed. The leading subjects will be dosed at intervals of at least 10 minutes, and the remaining subjects also at intervals of at least 10 minutes. To maintain the blind nature of the study, 1 of the leading subjects will be randomised to receive MGB-BP-3 and the other to placebo.

Part A is considered to be the 'first in human' portion of the study, so GP (General Practioner) replies must be obtained for the subjects in Part A. Subjects will be screened during the 4 weeks before their first dose of trial medication. In each of their 3 study sessions, subjects will be resident on the ward from the day before dosing (Day -1), until completion of procedures at 72 h after their dose of trial medication (Day 4). Subjects will attend a follow-up visit at 7-10 days after their dose of trial medication.

Part B Part B is a randomised, double-blind, placebo-controlled, sequential-group, repeated ascending-dose trial in 24 healthy men.

The sponsor and investigator will select 3 dose levels to be tested in Part B, based on available safety and tolerability data from Part A. The highest total daily dose tested in Part B will not exceed the highest dose in Part A that was acceptably tolerated and for which there were no safety concerns. Part B can start before Part A has finished, provided that the total daily dose to be given (or a higher dose) has previously been shown to be acceptably tolerated and safe in Part A.

Subjects will be enrolled in 3 groups of 8 (Groups 3-5). Each subject will have 1 study session, in which they will receive twice-daily oral doses of MGB-BP-3, or matching placebo, for 9 days (Days 1-9) and a single dose on the morning of Day 10.

In each group, 6 subjects will be randomised to receive MGB-BP-3 and 2 subjects will be randomised to receive placebo. Subjects in each group will be dosed at intervals of at least 10 minutes.

For each ascending dose level, there'll be a gap of least 6 days between the final dose of the previous group and the first dose of the next group. The investigator and sponsor will review safety and tolerability data for each dose level before increasing the dose. The dose will be escalated only if the safety and tolerability of the previous dose level are acceptable. The planned doses may be changed, depending on the safety and tolerability of previous doses - a dose level may be repeated or a lower dose tested.

Subjects will be screened within 4 weeks before their first dose of trial medication. They will be resident on the ward from admission on Day -2 until completion of procedures at 72 h after their final dose of trial medication (Day 13). They will attend a follow-up visit at 7-10 days after their final dose of trial medication.

Methods: Parts A and B

The following assessments will be made:

Safety: laboratory assessments (routine haematology, biochemistry and urinalysis), physical examination, 12-lead ECG, telemetry (Part A only) faecal occult blood, intestinal permeability (the ratio of lactulose to mannitol excreted in urine, Part B only), faecal flora (Part B only), vital signs, and adverse events.

Tolerability: adverse events. Pharmacokinetic: blood samples for assay of MGB-BP-3 and possible metabolites will be taken before, and frequently up to 48 h after dosing in Part A, and up to 12 h after subjects' morning dose on Day 1 and up to 48 h after dosing on Day 10 in Part B. In addition, in Part B, a blood sample will be taken before the morning dose on each of Days 2-9. Urine will be collected for 24 h after each dose for assay of MGB-BP-3 in Part A, and for 12 h after the morning dose on Day 1 and 10 (Part B only). Faecal samples will be collected daily until 72 h after subjects' (final) dose for assay of MGB-BP-3 in each study session, and in Part B for 24 h after dosing on Days 1 and 5.

Primary variables Safety: vital signs, ECG, telemetry (Part A only), physical examination, laboratory safety tests, faecal occult blood, intestinal permeability (Part B only), faecal flora (Part B only) Tolerability: adverse events

Secondary variables

Pharmacokinetics: PK parameters of MGB-BP-3:

Cmax, tmax and if appropriate t½, AUC0-t, AUC0-∞, Ctrough, AUC 0-τ (Part B), Vd/f (in Part A and Vdss/f in Part B) and CL/f (in Part A and CLss/f in Part B) in plasma Ae0-24 (Part A), Ae0-τ (Part B) and CLr in urine The amount of MGB-BP-3 excreted in faeces.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Body mass index (BMI) of 18.0-30.9 kg/m2
* Normal blood pressure
* healthy on the basis of a clinical history & physical examination
* Normal ECG
* Normal vital signs
* Normal laboratory tests of blood and urine
* Willing to use reliable contraception
* Able to give fully informed written consent

Exclusion Criteria:

* Positive tests for hepatitis B & C
* Positive tests for HIV
* Severe adverse reaction to any drug
* Drug or alcohol abuse
* Smoke more than 5 cigarettes (or use of equivalent tobacco or nicotine products) daily
* Received over-the-counter medication within previous 7 days (with the exception of paracetamol)
* Prescribed medication during previous 28 days
* Participation in other clinical trials of unlicensed medicines
* Loss of more than 400 mL blood, within the previous 3 months
* Vital signs outside the acceptable range
* Clinically relevant abnormal findings at the screening assessment
* Acute or chronic illness
* Clinically relevant abnormal medical history or concurrent medical condition
* Possibility that volunteer will not cooperate.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-07; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of single and repeated oral doses of MGB-BP-3 in healthy men | 4 months
  Safety Assessment - Composite Metrics: vital signs, ECG, telemetry (Part A only), physical examination, laboratory safety tests, faecal occult blood, intestinal permeability (absorptive capacity test using differential sugar absorption with the urine sugars measured using LC-MS, Part B only), faecal flora (Part B only) and Tolerability (AE's & SAE's)

SECONDARY OUTCOMES:
To assess the pharmacokinetics (PK) of single and repeated oral doses of MGB-BP-3 in healthy men | 4 months
  PK parameters of MGB-BP-3 - Composite Metrics Cmax, tmax and if appropriate t½, AUC0-t, AUC0-∞, Ctrough, AUC 0-τ (Part B), Vd/f (in Part A and Vdss/f in Part B) and CL/f (in Part A and CLss/f in Part B) in plasma Ae0-24 (Part A), Ae0-τ (Part B) and CLr in urine The amount of MGB-BP-3 excreted in faeces.

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Boyce, Various, Principal Investigator — HMR London

REFERENCES:
- See also: MGB Biopharma Limited — http://www.mgb-biopharma.com